CLINICAL TRIAL: NCT05705583
Title: A Companion Diagnostic Study to Develop Circulating Exosomes as Predictive Biomarkers for the Response to Immunotherapy in Renal Cell Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, ZHAO An, Zhejiang Cancer Hospital, Zhejiang Cancer Hospital
Other Study IDs: RCC-CDx-001
Record Dates: First submitted 2023-01-12; First posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Urine Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collection of blood and urine specimens from patients receiving immunotherapy as part of their standard of care for the treatment of RCC
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Other: Blood and Urine Collection — Blood and Urine Collection

SUMMARY:
Immune checkpoint inhibitors targeting PD-1 or PD-L1 have been developed and clinical trials showning better response in unselected patients with metastatic renal cell carcinoma (RCC). At the moment, no clear biomarker exists to accurately predict anti-PD1/PDL1 RCC responsiveness. The objective of this study is to develop and evaluate the utility of circulating exosomes as companion diagnostic biomarker for predicting response to immunotherapy in patients with RCC.

ELIGIBILITY:
Inclusion Criteria:

* Advanced Metastatic RCC
* Scheduled to initiate an immunocheckpoint inhibitors or in combination with them
* Age >= 18 years
* Able to provide informed consent

Exclusion Criteria:

* Other, unrelated, concomitant active, invasive malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with renal cell carcinoma
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The correlation between the circulating exosomes levels and the tumor responsiveness | 3 years
  The Measurement： The concentration of ciruculating exosomes and the expression level of exosomal RNA.
  The Measurement Tool:
  RT-PCR，WB and Elisa

CONTACTS AND LOCATIONS:
Locations (1):
- An Zhao, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang H, Zhu Z, Zhang Y, Jiang T, Zhang M, Wang Z, Zhang Y, Zhao A, Su B. New insight into immune checkpoint inhibitors in the treatment of advanced renal cell carcinoma. Sci China Life Sci. 2023 Apr;66(4):875-878. doi: 10.1007/s11427-022-2197-7. Epub 2022 Dec 1. No abstract available. PMID 36469217
- [Result] Yu M, Liu X, Xu H, Shen S, Wang F, Chen D, Li G, Wang Z, Zuo Z, Zhao A. Comprehensive Evaluation of the m6A Regulator Prognostic Risk Score in the Prediction of Immunotherapy Response in Clear Cell Renal Cell Carcinoma. Front Immunol. 2022 Jun 17;13:818120. doi: 10.3389/fimmu.2022.818120. eCollection 2022. PMID 35784363
- [Result] Zhang W, Ni M, Su Y, Wang H, Zhu S, Zhao A, Li G. MicroRNAs in Serum Exosomes as Potential Biomarkers in Clear-cell Renal Cell Carcinoma. Eur Urol Focus. 2018 Apr;4(3):412-419. doi: 10.1016/j.euf.2016.09.007. Epub 2016 Oct 14. PMID 28753793